CLINICAL TRIAL: NCT02317315
Title: Non-Invasive Sampling of Inflammatory Mediators Associated With Spontaneous Preterm Birth Less Than 32 Weeks Gestation
Brief Title: Biomarkers Associated With Spontaneous Preterm Birth Less Than 32 Wks Gestation
Status: Completed | Type: Observational
Sponsor: Ranjith Kamity, MD (Other)
Responsible Party: Sponsor-Investigator, Ranjith Kamity, MD, Principal Investigator, Winthrop University Hospital
Organization: Winthrop University Hospital (Other)
Other Study IDs: WinthropUH
Record Dates: First submitted 2014-12-10; First posted 2014-12-16 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Preterm Labor; Preterm Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Saliva - We will collect saliva in a sterile container.
  2. Maternal Blood - Blood samples will be collected during routine blood draws and into serum separator tubes, spun, and the serum stored at -80°C.
  3. Urine - Urine samples will be collected into a sterile container.
  4. Cervical and vaginal secretions - During speculum exam, we will simultaneously insert two Weck-Cell Sponges directly into the cervical os for collection of cervical secretions then another two sponges will be applied in the posterior fornix for collection of vaginal fluid.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm labor group: Patients who are admitted for evaluation of preterm labor.

SUMMARY:
Preterm delivery (PTD) is a leading cause of neonatal mortality and continues to be a major public health concern, reaching 12.9% in 2006, despite intense research to reverse this trend. Currently, fetal fibronectin (fFN) screening and cervical length determined by ultrasound are two tests which are proven to have benefit in the identification of those at greatest risk for preterm delivery. However the benefit of these tests is limited to situations where a negative result can avoid unnecessary interventions. Currently, maternal fetal monitoring is limited, as it is difficult to "see" what is going on in the placenta (maternal-fetal interface) without invasive measures such as placental biopsy or amniocentesis. Our goal for this study is to identify a group of biomarkers in non-invasive compartments (such as saliva, blood, urine, and/or cervical and vaginal secretions) that are associated with preterm labor and birth. We hypothesize that preterm labor will display an inflammatory profile, which consists of unique inflammatory biomarkers from different non-invasive bodily fluid compartments (such as Il-10 in urine, VEGF in cervical secretions, and IP-10 in saliva), that correlates with a high incidence of preterm birth.

DETAILED DESCRIPTION:
Preterm delivery (PTD) is a leading cause of neonatal mortality and continues to be a major public health concern, reaching 12.9% in 2006, despite intense research to reverse this trend. Currently, fetal fibronectin (fFN) screening and cervical length determined by ultrasound are two tests which are proven to have benefit in the identification of those at greatest risk for preterm delivery. However the benefit of these tests is limited to situations where a negative result can avoid unnecessary interventions. The first goal of this study is to identify non-invasive predictor(s) that will increase the clinician's ability to identify patients who present with second trimester preterm labor (PTL) at risk for preterm delivery (PTD) ≤ 32 weeks gestation.

Currently, maternal fetal monitoring is limited, as it is difficult to "see" what is going on in the placenta (maternal-fetal interface) without invasive measures such as placental biopsy or amniocentesis. Our preliminary study from term pregnancies has shown that a specific correlation of an intrauterine cytokine may be reflected in one noninvasive site but not another, depending upon the type of cytokine and the compartment from which it is secreted. Therefore, our second goal for this study is to identify inflammatory markers in non-invasive maternal compartments (such as saliva, blood, urine, and/or cervical and vaginal secretions) that have a strong association with placenta/fetal membranes at the time of preterm birth ≤ 32 weeks gestation.

Pregnant women, under 32 weeks gestation, who are admitted to Winthrop University Hospital for evaluation of preterm labor will be eligible for this study. Women with indicated preterm births (i.e. pre-eclampsia), multiple pregnancies, known major fetal abnormality (ex. those that are known to be incompatible with life) and premature rupture of membranes will be excluded from this study. After consent is obtained, samples (blood, urine, saliva, vaginal, and cervical secretions) will be obtained and biomarkers will be identified using a Bio-Plex cytokine concentration assay. These women will than be followed until they deliver. Women who deliver after 32 weeks gestation will form our control group and women who deliver before 32 weeks gestation will form our preterm birth group. Concentration of the biomarkers in the various maternal-fetal compartments will be analyzed and compared between the two groups. For all women who delivery ≤ 32 weeks gestation, non-invasive samples will also be collected around delivery and these cytokine levels will be compared to placenta/fetal membranes to access how well non-invasive fluids reflect the intrauterine environment.

We hypothesize that preterm labor will display an inflammatory profile, which consists of unique inflammatory biomarkers from different non-invasive bodily fluid compartments (such as Il-10 in urine, VEGF in cervical secretions, and IP-10 in saliva), that correlates with a high incidence of preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18-40 years old between 20 to 32 weeks gestation with singleton pregnancies and are admitted to Winthrop University Hospital for evaluation of preterm labor. Preterm labor will be defined as contractions every 5 minutes associated with cervical changes or cervical dilatation > 2cm with 80% effacement. Subjects must have reliable dates confirmed by early ultrasound.

Exclusion Criteria:

* Indicated preterm births (i.e. pre-eclampsia), multiple pregnancies, known major fetal abnormality (ex. those that are known to be incompatible with life) and premature rupture of membranes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females between the age of 18-40 who present in preterm labor will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-01-02 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | Within 5 months of Preterm labor

CONTACTS AND LOCATIONS:
Overall Officials: RANJITH KAMITY, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hosptial, Mineola, New York, United States